CLINICAL TRIAL: NCT01684215
Title: A PHASE 1/2 STUDY OF THE EFFICACY, SAFETY, AND PHARMACOKINETICS OF ORAL PD-0332991, A CYCLIN-DEPENDENT KINASE 4 AND 6 (CDK4/6) INHIBITOR, AS SINGLE AGENT IN JAPANESE PATIENTS WITH ADVANCED SOLID TUMORS OR IN COMBINATION WITH LETROZOLE FOR THE FIRST-LINE TREATMENT OF POSTMENOPAUSAL JAPANESE PATIENTS WITH ER (+) HER2 (-) ADVANCED BREAST CANCER
Brief Title: A Study Of Oral Palbociclib (PD-0332991), A CDK4/6 Inhibitor, As Single Agent In Japanese Patients With Advanced Solid Tumors Or In Combination With Letrozole For The First-Line Treatment Of Postmenopausal Japanese Patients With ER (+) HER2 (-) Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A5481010
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Results first posted 2017-05-02 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Neoplasms; Breast Neoplasms
Keywords: Phase 1/2; PD-0332991; palbociclib; Cyclin Dependent Kinase 4/6 inhibitor; Japanese; solid tumors; breast cancer; A5481010
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — palbociclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single-agent PD-0332991 (Experimental): Phase 1 Part 1
  Interventions: Drug: PD-0332991
- PD-0332991 in combination with letrozole (Experimental): Phase 1 Part 2
  Interventions: Drug: PD-0332991; Drug: letrozole
- PD-0332991 with letrozole (Experimental): Phase 2
  Interventions: Drug: PD-0332991; Drug: letrozole

INTERVENTIONS:
Drug: PD-0332991 — PD-0332991 (100 mg or 125 mg) will be orally administered once a day for 3 weeks followed by 1 week off treatment, in the morning on an empty stomach. Dose reduction of PD-0332991 by one (100 mg) or two (75 mg) dose level is permitted depending on treatment related toxicity.
  Arms: Single-agent PD-0332991
Drug: PD-0332991 — PD-0332991, 125 mg, will be orally administered with food once a day for 3 weeks followed by 1 week off treatment. PD-0332991 will be administered once a day together with letrozole. Dose reduction of PD-0332991 by one (100 mg) or two (75 mg) dose level is permitted depending on treatment related toxicity.
  Arms: PD-0332991 in combination with letrozole
Drug: letrozole — Letrozole, 2.5 mg, will be orally administered once a day in continuous daily dosing together with PD-0332991. Dose reduction of letrozole is not permitted, but dosing interruptions for letrozole-related toxicity are allowed as per investigator's medical judgement.
  Arms: PD-0332991 in combination with letrozole
Drug: PD-0332991 — PD-0332991, 125 mg, will be orally administered with food once a day for 3 weeks followed by 1 week off treatment. PD-0332991 will be administered once a day together with letrozole. Dose reduction of PD-0332991 by one (100 mg) or two (75 mg) dose level is permitted depending on treatment related toxicity.
  Arms: PD-0332991 with letrozole
Drug: letrozole — Letrozole, 2.5 mg, will be orally administered once a day in continuous daily dosing together with PD-0332991. Dose reduction of letrozole is not permitted, but dosing interruptions for letrozole-related toxicity are allowed as per investigator's medical judgement.
  Arms: PD-0332991 with letrozole

SUMMARY:
This study is comprised of two portions: a Phase 1 portion and a Phase 2 portion. The Phase 1 portion is a single-country, non-randomized, open label, clinical trial which will evaluate the safety, tolerability, preliminary efficacy, and PK profile of PD-0332991 as a single agent in Japanese patients with advanced solid tumors, and PD-0332991 in combination with letrozole in the first-line treatment of Japanese patients with ER(+) HER2(-) ABC. The Phase 2 portion is a single-country, non-randomized, open-label, single-cohort, multi-center clinical trial to evaluate the efficacy and safety of PD-0332991 in combination with letrozole for the first-line treatment of postmenopausal Japanese patients with ER(+) HER2(-) ABC.

ELIGIBILITY:
Inclusion Criteria:

Phase 1

* In Part 1, advanced solid tumor (except SCLC or retinoblastoma) proven histologically or cytologically at original diagnosis, that is refractory to standard therapy or for whom no standard of care therapy is available.
* In Part 2 and Phase 2, post menopausal women with proven diagnosis of ER-positive, HER2-negative adenocarcinoma of the breast with evidence of locoregionally recurrent or metastatic disease (including bone only disease) not amenable to resection or radiation therapy with curative intent and for whom chemotherapy is not clinically indicated.
* Adequate blood cell counts, kidney function and liver function and and Eastern Cooperative Oncology Group [ECOG] score of 0 or 1.
* Resolved acute effects of any prior therapy to baseline severity or Grade ≤1

Phase 2

* Adult women (≥ 20 years of age) with proven diagnosis of adenocarcinoma of the breast with evidence of locoregionally recurrent or metastatic disease not amenable to resection or radiation therapy with curative intent and for whom chemotherapy is not clinically indicated.
* Documentation of histologically or cytologically confirmed diagnosis of ER(+) breast cancer based on local laboratory results.
* Adequate blood cell counts, kidney function and liver function and and Eastern Cooperative Oncology Group [ECOG] score of 0 to 2.

Exclusion Criteria:

Phase 1

* Active uncontrolled or symptomatic CNS metastases.
* Uncontrolled infection, unstable or sever intercurrent medical condition, or current drug or alcohol abuse
* Active or unstable cardiac disease or history of heart attack within 6 months

Phase 2

* HER2 positive tumor based on local laboratory results utilizing one of the sponsor approved assays.
* Known active uncontrolled or symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease.
* Prior neoadjuvant or adjuvant treatment with a non steroidal aromatase inhibitor (ie, anastrozole or letrozole) with disease recurrence while on or within 12 months of completing treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-10-19 (Actual); Primary Completion 2016-03-04 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- Japan (16):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kumamoto Shinto General Hospital, Kumamoto, Kumamoto
  - Saitama Cancer Center, Kita-adachi-gun, Saitama
  - National Cancer Center Hospital, Chuo-Ku, Tokyo
  - Chiba Cancer Center, Chiba
  - National Hospital Organization Shikoku Cancer Center, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Hakuaikai Medical Corporation Sagara Hospital, Kagoshima
  - Kumamoto University Hospital, Kumamoto
  - Kumamoto City Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Iwate Medical University Hospital, Numakunai
  - National Hospital Organization Osaka National Hospital, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Takahashi M, Masuda N, Nishimura R, Inoue K, Ohno S, Iwata H, Hashigaki S, Muramatsu Y, Umeyama Y, Toi M. Palbociclib-letrozole as first-line treatment for advanced breast cancer: Updated results from a Japanese phase 2 study. Cancer Med. 2020 Jul;9(14):4929-4940. doi: 10.1002/cam4.3091. Epub 2020 May 18. PMID 32420697
- [Derived] Masuda N, Mukai H, Inoue K, Rai Y, Ohno S, Mori Y, Hashigaki S, Muramatsu Y, Umeyama Y, Iwata H, Toi M. Neutropenia management with palbociclib in Japanese patients with advanced breast cancer. Breast Cancer. 2019 Sep;26(5):637-650. doi: 10.1007/s12282-019-00970-7. Epub 2019 May 24. PMID 31127500
- [Derived] Tamura K, Mukai H, Naito Y, Yonemori K, Kodaira M, Tanabe Y, Yamamoto N, Osera S, Sasaki M, Mori Y, Hashigaki S, Nagasawa T, Umeyama Y, Yoshino T. Phase I study of palbociclib, a cyclin-dependent kinase 4/6 inhibitor, in Japanese patients. Cancer Sci. 2016 Jun;107(6):755-63. doi: 10.1111/cas.12932. Epub 2016 May 11. PMID 26991823
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481010&StudyName=A%20Study%20Of%20Oral%20Palbociclib%20%28PD-0332991%29%2C%20A%20CDK4/6%20Inhibitor%2C%20As%20Single%20Agent%20In%20Japanese%20Patients%20With%20Advanced%20Solid%20Tumors%20Or

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study comprised of 2 phases: Participants were enrolled to dose escalation cohorts (PD-0332991 100 milligram [mg] and 125 mg) in Phase 1 Part 1, to maximum tolerated dose (MTD) cohort (PD-0332991 125 mg+ Letrozole 2.5 mg) in Phase 1 Part 2 and to expanded cohort (PD-0332991 125 mg and Letrozole 2.5 mg) in Phase 2.
Groups:
- PD-0332991 100 mg: Dose Escalation Cohort: In Phase 1-Part 1, participants received single oral dose of PD-0332991 100 mg capsule in lead-in period (7 days prior to Cycle 1 Day 1), followed by PD-0332991 100 mg capsule orally once daily continuously for 21 days followed by 7 days off treatment in each cycle of 28 days, unless participants experienced disease progression or unacceptable toxicity or withdrew consent.
- PD-0332991 125 mg: Dose Escalation Cohort: In Phase 1-Part 1, participants received single oral dose of PD-0332991 125 mg capsule in lead-in period (7 days prior to Cycle 1 Day 1), followed by PD-0332991 125 mg capsule orally once daily continuously for 21 days followed by 7 days off treatment in each cycle of 28 days, unless participants experienced disease progression or unacceptable toxicity or withdrew consent.
- PD-0332991 125 mg+ Letrozole 2.5 mg: MTD Cohort: In Phase1-Part 2, participants received Letrozole 2.5 mg tablet along with PD-0332991 125 mg capsule orally once daily continuously for 21 days followed by 7 days off treatment in each cycle of 28 days, unless participants experienced disease progression or unacceptable toxicity or withdrew consent.
- PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort: In Phase 2, participants received Letrozole 2.5 mg tablet along with PD-0332991 125 mg capsule orally once daily continuously for 21 days followed by 7 days off treatment in each cycle of 28 days, unless participants experienced disease progression or unacceptable toxicity or withdrew consent.
Period: Phase 1, Part 1
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort | PD-0332991 125 mg+ Letrozole 2.5 mg: MTD Cohort | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Started | 6 | 6 | 0 | 0
Treated | 6 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Objective progression or relapse | 5 | 6 | 0 | 0
Period: Phase 1, Part 2
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort | PD-0332991 125 mg+ Letrozole 2.5 mg: MTD Cohort | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Started | 0 | 0 | 6 (Eligible participants who consented for Phase 1 Part 2.) | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 6 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Commercial avaliabity of Palbociclib | 0 | 0 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Phase 2
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort | PD-0332991 125 mg+ Letrozole 2.5 mg: MTD Cohort | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Started | 0 | 0 | 0 | 43 (Eligible participants who consented for Phase 2.)
Treated | 0 | 0 | 0 | 42
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 43
Not completed — Death | 0 | 0 | 0 | 8
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 30
Not completed — Enrolled but not treated | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991).
Groups:
- Total: Total of all reporting groups
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort | PD-0332991 125 mg+ Letrozole 2.5 mg: MTD Cohort | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort | Total
Number analyzed (Participants) | 6 | 6 | 6 | 42 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 4 | 26 | 39
  >=65 years | 2 | 1 | 2 | 16 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 6 | 42 | 55
  Male | 1 | 4 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLT): Part 1 Phase 1
Description: DLT was classified as per common terminology criteria for adverse events (CTCAE) version 4.0 as any of the events occurring during 28 days of Cycle 1,attributed to study drug:grade 4 neutropenia(for a duration of greater than [>]7 days); febrile neutropenia (grade greater than or equal to [>=]3 neutropenia,body temperature >=38.5 degree Celsius);grade >=3 thrombocytopenia with bleeding episode;grade 4 thrombocytopenia;grade >=3 non-hematologic toxicity except grade 3 or more nausea, vomiting,electrolyte abnormality(if controllable by therapy);grade 3 QTc prolongation(>500 millisecond [msec])persist after correction of reversible cause such as electrolyte abnormalities or hypoxia. Lack of hematologic recovery (platelets less than [<]50,000/microliter [mcL],absolute neutrophil count <1,000/mcL,hemoglobin <8.0 gram/deciliter [g/dL]) or prolonged non hematologic toxicities that delays initiation of next dose by >7 days;receipt of <75 percent of planned dose in first cycle due to toxicity.
Time Frame: Lead-in period (Day -7) up to Day 28 (Cycle 1)
Population: DLT analysis set included all participants whom DLTs were evaluable in Part 1 Phase 1.
Measure: Count of Participants; unit: Participants
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
Participants | 1 | 1

2. Primary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs): Part 2 Phase 1
Description: A treatment related AE is any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event had a causal relationship with the treatment or usage. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
  Relatedness was judged by investigator. AEs included both serious and non-serious adverse events.
Time Frame: Baseline (Day 1) up to 28 days after last dose of study drug (up to 1673 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991).
Measure: Count of Participants; unit: Participants
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: MTD Cohort
Number analyzed (Participants) | 6
Participants
  AEs | 6
  SAEs | 2

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) By Severity: Part 2 Phase 1
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An AE was considered treatment emergent if occurred for the first time after the start of study treatment or occurred prior to the start of treatment but increased in National Cancer Institute (NCI) CTCAE grade during study treatment period. AE severity was defined to be the maximum toxicity grade of the TEAEs experienced by the participants during the study. AE was assessed according to severity as: Grade 1 (mild AE), Grade 2 (moderate AE), Grade 3 (severe AE), Grade 4 (life-threatening consequences) and Grade 5 (death related to AE).
Time Frame: Baseline (Day 1) up to 28 days after last dose of study drug (up to 1673 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991).
Measure: Count of Participants; unit: Participants
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: MTD Cohort
Number analyzed (Participants) | 6
Participants
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 4
  Grade 4 | 2
  Grade 5 | 0

4. Primary Outcome: Percentage of Participants With 1 Year Progression Free Survival (PFS): Phase 2
Description: PFS was defined as the time from first dose of study treatment to the date of the first documentation of objective progression of disease (PD) or death due to any cause in the absence of documented PD, whichever occurred first. PD was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.1-year PFS was defined as the percentage of participants without PFS events (PD or death due to any cause) at 12 months based on the Kaplan-Meier estimate. Percentage of participants with 1-year PFS with 90% confidence interval (CI) were reported.
Time Frame: From initiation of treatment up to 12 months
Population: Full analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991).
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 42
percentage of participants | 75.6 [62.4 to 84.7]

5. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs): Phase 1 (Part 1) and Phase 2
Description: as for outcome 2
Time Frame: Part 1 Phase 1: Lead-in period (Day -7) up to 28 days after last dose of study drug (up to 308 days), Phase 2: Baseline (Day 1) up to 28 days after last dose of study drug (up to 1526 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991).
Measure: Count of Participants; unit: Participants
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 6 | 6 | 42
Participants
  AEs | 6 | 5 | 42
  SAEs | 0 | 0 | 2

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) By Severity: Phase 1 (Part 1) and Phase 2
Description: AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An AE was considered treatment emergent if occurred for the first time after the start of study treatment or occurred prior to the start of treatment but increased in NCI CTCAE version 4.0 grade during study treatment period. AE severity was defined to be the maximum toxicity grade of the TEAEs experienced by the participants during the study. AE was assessed according to severity as: Grade 1 (mild AE), Grade 2 (moderate AE), Grade 3 (severe AE), Grade 4 (life-threatening consequences) and Grade 5 (death related to AE).
Time Frame: as for outcome 5
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991).
Measure: Count of Participants; unit: Participants
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 6 | 6 | 42
Participants
  Grade 1 | 0 | 1 | 0
  Grade 2 | 0 | 1 | 2
  Grade 3 | 4 | 3 | 29
  Grade 4 | 2 | 1 | 10
  Grade 5 | 0 | 0 | 1

7. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Abnormality criteria: hemoglobin: <0.8*lower limit of normal [LLN], platelets: <0.5*LLN or >1.75*upper limit of normal [ULN], leukocytes: <0.6*LLN or >1.5*ULN, lymphocytes, total neutrophils: <0.8*LLN or >1.2*ULN, basophils, eosinophil,monocytes: >1.2*ULN); aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma glutamyl transferase (GT): >0.3*ULN, total protein, albumin: <0.8*LLN or >1.2*ULN, total bilirubin, direct bilirubin: >1.5*ULN; blood urea nitrogen, creatinine: >1.3*ULN, uric acid: >1.2*ULN; sodium: <0.95*LLN or >1.05*ULN, potassium, chloride, calcium, magnesium: <0.9*LLN or >1.1*ULN, phosphate: <0.8*LLN or >1.2*ULN; creatine kinase: >2.0*ULN, glucose fasting: <0.6*LLN or >1.5*ULN, glycosylated haemoglobin: >1.3*ULN;urinalysis dipstick (urine protein, urine blood >=1); urine protein 24 hour: >1.1*ULN; coagulation Activated partial thromboplastin time [APTT], Prothrombin, prothrombin international ratio: >1.1*ULN.
Time Frame: Part 1 Phase 1: Lead-in period (Day -7) up to 308 days; Part 2 Phase 1: Baseline (Day 1) up to 1673 days; Phase 2: Baseline (Day 1) up to 1526 days
Population: Safety analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991).
Measure: Count of Participants; unit: Participants
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort | PD-0332991 125 mg+ Letrozole 2.5 mg: MTD Cohort | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 42
Participants | 6 | 6 | 6 | 40

8. Secondary Outcome: Area Under the Plasma Concentration Time Curve Over Dosing Interval (AUCtau) of PD-0332991 Following Multiple Dose: Part 1 Phase 1
Description: AUCtau is area under the plasma concentration-time curve over dosing interval which is calculated by log-linear trapezoidal method.
Time Frame: Multiple dose: 0 hour (pre-dose), 1, 2, 4, 6, 8, 12, 24 hours post-dose on Cycle 1 Day 8
Population: Pharmacokinetic (PK) parameter analysis set included treated participants who had at least 1 of the PK parameters of primary interest in at least 1 PK sampling period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
nanogram*hour per milliliter (ng*hr/mL) | 1276 (45) | 2838 (43)

9. Secondary Outcome: AUCtau Dose Normalized to 125 Milligram (mg) of PD-0332991 Following Multiple Dose: Part 1 Phase 1
Description: AUCtau Dose Normalized to 125 mg is area under the plasma concentration-time curve over dosing interval dose normalized to 125 mg which is calculated by log-linear trapezoidal method.
Time Frame: Multiple dose: 0 hour (pre-dose), 1, 2, 4, 6, 8, 12, 24 hours post-dose on Cycle 1 Day 8
Population: PK parameter analysis set included treated participants who had at least 1 of the PK parameters of primary interest in at least 1 PK sampling period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 1595 (45) | 2838 (43)

10. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From 0 to Time 24 Hours (AUC24) of PD-0332991 Following Single Dose: Part 1 Phase 1
Description: AUC24 is area under the plasma concentration-time curve from 0 to time 24 hours which is calculated by log-linear trapezoidal method.
Time Frame: Single dose: 0 hour (pre-dose), 1, 2, 4, 6, 8, 12 and 24 hours post-dose in Lead-in period (Day -7)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 547.5 (19) | 1322 (42)

11. Secondary Outcome: AUC24 Dose Normalized to 125 mg of PD-0332991 Following Single Dose: Part 1 Phase 1
Description: AUC24 Dose Normalized to 125 mg is area under the plasma concentration-time curve from 0 to time 24 hours dose normalized to 125 mg which is calculated by log-linear trapezoidal method.
Time Frame: Single dose: 0 hour (pre-dose), 1, 2, 4, 6, 8, 12 and 24 hours post-dose in Lead-in period (Day -7)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 684.5 (19) | 1322 (42)

12. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUCinf) of PD-0332991 Following Single Dose: Part 1 Phase 1
Description: AUCinf is area under the plasma concentration-time curve from 0 to infinity which is calculated by log-linear trapezoidal method.
Time Frame: Single dose: 0 hour (pre-dose), 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose in Lead-in period (Day -7)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 1039 (32) | 2483 (49)

13. Secondary Outcome: AUCinf Dose Normalized to 125 mg of PD-0332991 Following Single Dose: Part 1 Phase 1
Description: AUCinf Dose Normalized to 125 mg is area under the plasma concentration-time curve from 0 to infinity dose normalized to 125 mg which is calculated by log-linear trapezoidal method.
Time Frame: Single dose: 0 hour (pre-dose), 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose in Lead-in period (Day -7)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 1296 (32) | 2483 (49)

14. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From 0 to Time of Last Measurable Concentration (AUClast) of PD-0332991 Following Single Dose: Part 1 Phase 1
Description: AUClast is area under the plasma concentration-time curve from 0 to time of last measurable concentration which is calculated by log-linear trapezoidal method.
Time Frame: Single dose: 0 hour (pre-dose), 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose in Lead-in period (Day -7)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 971.7 (31) | 2396 (48)

15. Secondary Outcome: AUClast Dose Normalized to 125 mg of PD-0332991 Following Single Dose: Part 1 Phase 1
Description: AUClast Dose Normalized to 125 mg is area under the plasma concentration-time curve from 0 to time of last measurable concentration dose normalized to 125 mg which is calculated by log-linear trapezoidal method.
Time Frame: Single dose: 0 hour (pre-dose), 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose in Lead-in period (Day -7)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 1215 (31) | 2396 (48)

16. Secondary Outcome: Apparent Oral Clearance of PD-0332991: Part 1 Phase 1
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. It was calculated by dividing the given oral dose by AUCinf. AUCinf is area under the plasma concentration-time curve from 0 to infinity which is calculated by log-linear trapezoidal method.
Time Frame: Single dose: 0 hour (pre-dose),1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose in Lead-in period (Day -7), Multiple dose: 0 hour (pre-dose), 1, 2, 4, 6, 8, 12, 24 hours post-dose on Cycle 1 Day 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
liter per hour (L/hr)
  Single dose | 96.43 (32) | 50.29 (49)
  Multiple dose | 78.43 (45) | 44.03 (43)

17. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Of PD-0332991: Part 1 Phase 1
Description: Cmax is maximum plasma concentration which is observed directly from the actual time-concentration data.
Time Frame: as for outcome 16
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
nanogram per milliliter (ng/mL)
  Single dose | 41.37 (15) | 104.1 (39)
  Multiple dose | 77.36 (33) | 185.5 (27)

18. Secondary Outcome: Cmax Dose Normalized to 125 mg of PD-0332991: Part 1 Phase 1
Description: Cmax Dose Normalized to 125 mg is maximum plasma concentration dose normalized to 125 mg which is observed directly from the actual time-concentration data.
Time Frame: as for outcome 16
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
ng/mL
  Single dose | 51.74 (15) | 104.1 (39)
  Multiple dose | 96.72 (33) | 185.5 (27)

19. Secondary Outcome: Pre-dose Plasma Concentration (Ctrough) of PD-0332991 Following Multiple Dose: Part 1 Phase 1
Description: Ctrough is pre-dose concentration during multiple dosing which is observed directly from the actual time-concentration data.
Time Frame: Multiple dose: 0 hour (pre-dose), 1, 2, 4, 6, 8, 12, 24 hours post-dose on Cycle 1 Day 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
ng/mL | 35.51 (59) | 72.76 (48)

20. Secondary Outcome: Accumulation Ratio (Rac) of PD-0332991 Following Multiple Dose: Part 1 Phase 1
Description: Rac is the ratio of AUCtau (after multiple doses) to AUCtau (after single dose). AUCtau is area under the plasma concentration-time curve over dosing interval which is calculated by log-linear trapezoidal method.
Time Frame: Single dose: 0 hour (pre-dose), 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose in Lead-in period (Day -7), Multiple dose: 0 hour (pre-dose), 1, 2, 4, 6, 8, 12, 24 hours post-dose on Cycle 1 Day 8
Population: as for outcome 9
Measure: Median (Full Range); unit: ratio
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
ratio | 2.060 [1.81 to 3.54] | 1.855 [1.74 to 3.10]

21. Secondary Outcome: Linearity (Rss) of PD-0332991 Following Multiple Dose: Part 1 Phase 1
Description: Rss is the ratio of AUCtau (after multiple doses) to AUCinf (after single dose). AUCtau is area under the plasma concentration-time curve over dosing interval which is calculated by log-linear trapezoidal method. AUCinf is area under the plasma concentration-time curve from 0 to infinity which is calculated by log-linear trapezoidal method.
Time Frame: as for outcome 20
Population: as for outcome 9
Measure: Median (Full Range); unit: ratio
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
ratio | 1.130 [1.03 to 1.73] | 1.105 [0.851 to 1.51]

22. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PD-0332991: Part 1 Phase 1
Description: Tmax is time at which maximum plasma concentration (Cmax) was observed. It was observed directly from data as time of first occurrence.
Time Frame: as for outcome 16
Population: as for outcome 9
Measure: Median (Full Range); unit: hour
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
hour
  Single dose | 5.02 [3.97 to 8.02] | 4.00 [3.90 to 8.00]
  Multiple dose | 4.02 [3.97 to 6.00] | 4.02 [3.95 to 6.02]

23. Secondary Outcome: Terminal Half-Life (t1/2) of PD-0332991: Part 1 Phase 1
Description: t1/2 is terminal elimination half-life which is calculated by loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: as for outcome 16
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
hour
  Single dose | 25.72 (5.2632) | 23.93 (2.6882)
  Multiple dose | 23.75 (6.7778) | 23.15 (7.7045)

24. Secondary Outcome: Volume of Distribution (Vz/F) of PD-0332991 Following Single Dose: Part 1 Phase 1
Description: Vz/F is apparent volume of distribution estimated from terminal phase, which is calculated as CL/F/kel. Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. It was calculated by dividing the given oral dose by area under the plasma concentration-time curve from 0 to infinity which is calculated by log-linear trapezoidal method (AUCinf). kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Single dose: 0 hour (pre-dose), 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose in Lead-in period (Day -7)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort
Number analyzed (Participants) | 6 | 6
liter | 3514 (25) | 1730 (41)

25. Secondary Outcome: Area Under the Plasma Concentration Time Curve Over Dosing Interval (AUCtau) of PD-0332991: Phase 2
Description: as for outcome 8
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post dose on Cycle 1 Day 15
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 6
ng*hr/mL | 1979 (16)

26. Secondary Outcome: Apparent Oral Clearance of PD-0332991: Phase 2
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. It was calculated by dividing the given oral dose by AUCtau. AUCtau is the area under the plasma concentration-time curve over dosing interval which is calculated by log-linear trapezoidal method.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post dose on Cycle 1 Day 15
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 6
L/hr | 63.21 (16)

27. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) Of PD-0332991: Phase 2
Description: Cmax is maximum plasma concentration which is observed directly from the actual time-concentration data.
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post dose on Cycle 1 Day 15
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 6
ng/mL | 124.7 (26)

28. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PD-0332991: Phase 2
Description: as for outcome 22
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post dose on Cycle 1 Day 15
Population: as for outcome 9
Measure: Median (Full Range); unit: hour
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 6
hour | 4.90 [2.00 to 8.20]

29. Secondary Outcome: Pre-dose Plasma Concentration (Ctrough) of PD-0332991: Phase 2
Description: as for outcome 19
Time Frame: 0 (pre-dose), 1, 2, 4, 6, 8, 10, 24 hours post dose on Cycle 1 Day 15
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 6
ng/mL | 59.75 (38)

30. Secondary Outcome: Percentage of Participants With Objective Response: Phase 1
Description: Objective response (OR) was defined as a complete response (CR) or partial response (PR) according to the RECIST version 1.1 recorded from first dose of study treatment until disease progression or death due to any cause. CR was defined as disappearance of all target lesions with the exception of nodal disease. All target nodes reduced to normal size (short axis <10 millimeter [mm]). PR was defined as a >=30 percent decrease in sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions. Percentage of participants with objective response (who achieved CR or PR) were reported.
Time Frame: From initiation of treatment up to disease progression (up to 30 months)
Population: Full analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991).
Measure: Number; unit: percentage of participants
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort | PD-0332991 125 mg+ Letrozole 2.5 mg: MTD Cohort
Number analyzed (Participants) | 6 | 6 | 6
percentage of participants
  With Complete Response | 0 | 0 | 0
  With Partial Response | 0 | 0 | 33.3

31. Secondary Outcome: Percentage of Participants With Objective Response: Phase 2
Description: Objective response was defined as a complete response (CR) or partial response (PR) according to the RECIST version 1.1 recorded from first dose of study treatment until disease progression or death due to any cause. PD was defined using RECIST v1.1, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. CR was defined as disappearance of all target lesions with the exception of nodal disease. All target nodes reduced to normal size (short axis <10 mm). PR was defined as a >=30% decrease in sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions. Percentage of participants with objective response (who achieved CR or PR) were reported.
Time Frame: From initiation of treatment up to disease progression (up to 1526 days)
Population: Full analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991).
Measure: Number; unit: percentage of participants
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 42
percentage of participants | 47.6

32. Secondary Outcome: Duration of Response (DOR): Part 2 Phase 1
Description: Duration of response was defined as the interval from the first documentation of objective tumor response in participants with CR (disappearance of all target lesions with the exception of nodal disease. All target nodes reduced to normal size (short axis <10 millimeter [mm]) or PR (a >=30 percent decrease in sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions) according to RECIST version 1.1 to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first.
Time Frame: baseline up to 1673 days
Population: Full analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991). Data for this outcome measure was not summarized and individual participant's data was reported. Here, number of participants analyzed (N) signifies the participants evaluable for this outcome measure.
Measure: Number; unit: days
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: MTD Cohort
Number analyzed (Participants) | 2
days
  Participant 1 | 1509
  Participant 2 | 1428

33. Secondary Outcome: Duration of Response (DOR): Phase 2
Description: Duration of response was defined as the interval from the first documentation of objective tumor response in participants with CR (disappearance of all target lesions with the exception of nodal disease, all target nodes reduced to normal size (short axis <10 mm) or PR (a >=30 % decrease in sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions) according to RECIST version 1.1 to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first. PD was defined using RECIST v1.1, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From initiation of treatment up to disease progression (up to 1526 days)
Population: Full analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991). Here, "Overall Number of Participants Analyzed" (N) signifies the participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 20
months | 41.4 [19.0 to NA] — Due to low number of participants with disease progression, upper limit of 95% confidence interval (CI) was not reached.

34. Secondary Outcome: Progression Free Survival (PFS): Part 2 Phase 1
Description: PFS was defined as the time from first dose of study treatment to the date of the first documentation of objective progression of disease (PD) or death due to any cause in the absence of documented PD, whichever occurs first. PD was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: baseline up to 1673 days
Population: Full analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991). Data for this outcome measure was not summarized and individual participant's data was reported.
Measure: Number; unit: days
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: MTD Cohort
Number analyzed (Participants) | 6
days
  Participant 1 | 1590
  Participant 2 | 1593
  Participant 3 | 1602
  Participant 4 | 36
  Participant 5 | 31
  Participant 6 | 1512

35. Secondary Outcome: Percentage of Participants With Disease Control (DC): Phase 2
Description: DC: CR, PR or stable disease (SD) for >=24 weeks according to RECIST version (v)1.1 recorded in time period between first dose of study treatment and disease progression or death to any cause. CR: disappearance of all target lesions with exception of nodal disease. All target nodes reduced to normal size (short axis <10 mm). PR: >=30% decrease in sum of longest dimensions of target lesions taking as a reference baseline sum longest dimensions. SD was defined as not achieving an OR with confirmed CR or PR according to RECIST v1.1, as determined by investigators, relative to response evaluable population, but remained stable for at least 24 weeks after first dose, then best overall response for such a participant was considered as stable disease. PD was defined using RECIST v1.1 as a 20% increase in sum of longest diameter of target lesions, or a measurable increase in a non-target lesion, or appearance of new lesions.
Time Frame: From initiation of treatment up to disease progression (up to 1526 days)
Population: Full analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991).
Measure: Number; unit: percentage of participants
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 42
percentage of participants | 85.7

36. Secondary Outcome: Overall Survival (OS): Phase 2
Description: Overall survival was defined as the time from first dose of study treatment to date of death due to any cause. In the absence of confirmation of death, survival time was censored to last date the participant was known to be alive. OS was estimated with Kaplan-Meier method.
Time Frame: From initiation of treatment up to follow-up period (up to 1526 days)
Population: Full analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 42
months | NA [47.5 to NA] — Due to low number of participants with event, median and upper limit of 95% CI was not reached.

37. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B): Phase 2 at Day 1 of Cycle 2, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, 35, 37, 39, 41, 43, 45, 47, 49 and End of Treatment
Description: The functional assessment of cancer therapy (FACT) is a modular approach to assess participant's health-related quality of life. FACT-B total score was derived from the sum of these 5 sub-scale scores: physical well-being, social/family well-being and functional well-being (all 3 sub-scales consisting of 7 items ranging from 0 to 28, where higher scores indicating better quality of life), emotional well-being (consists of 6 items and ranging from 0 to 24, where higher scores indicating better quality of life, and a breast cancer subscale (consists of 9 items and ranging from 0 to 36, where higher scores indicating better quality of life). Each individual item was rated on a 5-point Likert scale, ranging from 0 (not at all good) to 4 (very well), where higher scores indicating better quality of life. FACT-B total score range was of 0 (not at all good) to 144 (very well), where higher scores indicating better quality of life.
Time Frame: Baseline (Day 1 of Cycle 1), Day 1 of Cycle 2, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, 35, 37, 39, 41, 43, 45, 47, 49, End of treatment (up to 1526 days)
Population: Patient reported outcome (PRO) analysis set included all enrolled participants who receive at least 1 dose of study drug with both baseline and at least 1 complete post-baseline PRO assessment. "Number analyzed" signifies number of participants evaluable for specified time points.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 42
units on a scale
  Baseline | 106.46 [101.87 to 111.04]
  Change at Cycle 2: Day 1 | -1.20 [-4.56 to 2.16]
  Change at Cycle 3: Day 1: number analyzed (Participants) | 41
  Change at Cycle 3: Day 1 | -2.22 [-6.27 to 1.83]
  Change at Cycle 5: Day 1: number analyzed (Participants) | 38
  Change at Cycle 5: Day 1 | -2.38 [-6.07 to 1.31]
  Change at Cycle 7: Day 1: number analyzed (Participants) | 35
  Change at Cycle 7: Day 1 | -4.62 [-8.43 to -0.81]
  Change at Cycle 9: Day 1: number analyzed (Participants) | 35
  Change at Cycle 9: Day 1 | -4.45 [-7.86 to -1.04]
  Change at Cycle 11: Day 1: number analyzed (Participants) | 33
  Change at Cycle 11: Day 1 | -4.48 [-7.99 to -0.97]
  Change at Cycle 13: Day 1: number analyzed (Participants) | 29
  Change at Cycle 13: Day 1 | -6.32 [-10.56 to -2.09]
  Change at Cycle 15: Day 1: number analyzed (Participants) | 28
  Change at Cycle 15: Day 1 | -4.06 [-7.84 to -0.27]
  Change at Cycle 17: Day 1: number analyzed (Participants) | 28
  Change at Cycle 17: Day 1 | -6.07 [-9.48 to -2.65]
  Change at Cycle 19: Day 1: number analyzed (Participants) | 27
  Change at Cycle 19: Day 1 | -7.39 [-12.06 to -2.72]
  Change at Cycle 21: Day 1: number analyzed (Participants) | 27
  Change at Cycle 21: Day 1 | -5.85 [-10.29 to -1.42]
  Change at Cycle 23: Day 1: number analyzed (Participants) | 26
  Change at Cycle 23: Day 1 | -5.89 [-10.97 to -0.82]
  Change at Cycle 25: Day 1: number analyzed (Participants) | 24
  Change at Cycle 25: Day 1 | -4.22 [-8.61 to 0.17]
  Change at Cycle 27: Day 1: number analyzed (Participants) | 24
  Change at Cycle 27: Day 1 | -4.76 [-9.22 to -0.30]
  Change at Cycle 29: Day 1: number analyzed (Participants) | 23
  Change at Cycle 29: Day 1 | -6.26 [-10.94 to -1.57]
  Change at Cycle 31: Day 1: number analyzed (Participants) | 21
  Change at Cycle 31: Day 1 | -5.13 [-9.46 to -0.79]
  Change at Cycle 33: Day 1: number analyzed (Participants) | 20
  Change at Cycle 33: Day 1 | -7.12 [-11.14 to -3.11]
  Change at Cycle 35: Day 1: number analyzed (Participants) | 20
  Change at Cycle 35: Day 1 | -7.68 [-11.66 to -3.70]
  Change at Cycle 37: Day 1: number analyzed (Participants) | 19
  Change at Cycle 37: Day 1 | -8.07 [-12.56 to -3.58]
  Change at Cycle 39: Day 1: number analyzed (Participants) | 15
  Change at Cycle 39: Day 1 | -6.87 [-10.89 to -2.85]
  Change at Cycle 41: Day 1: number analyzed (Participants) | 11
  Change at Cycle 41: Day 1 | -5.70 [-11.41 to 0.02]
  Change at Cycle 43: Day 1: number analyzed (Participants) | 6
  Change at Cycle 43: Day 1 | -10.42 [-17.24 to -3.59]
  Change at Cycle 45: Day 1: number analyzed (Participants) | 3
  Change at Cycle 45: Day 1 | -7.94 [-26.09 to 10.20]
  Change at Cycle 47: Day 1: number analyzed (Participants) | 3
  Change at Cycle 47: Day 1 | -8.56 [-22.48 to 5.36]
  Change at Cycle 49: Day 1: number analyzed (Participants) | 2
  Change at Cycle 49: Day 1 | -10.58 [-66.70 to 45.54]
  End of Treatment: number analyzed (Participants) | 39
  End of Treatment | -9.17 [-13.82 to -4.52]

38. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-General (FACT-G): Phase 2 at Day 1 of Cycle 2, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, 35, 37, 39, 41, 43, 45, 47, 49 and End of Treatment
Description: FACT is a modular approach to assess participant's health-related quality of life. FACT-G total score was derived from the sum of these 4 sub-scale scores: physical well-being, social/family well-being and functional well-being (all 3 sub-scales consisting of 7 items ranging from 0 to 28, where higher scores indicating better quality of life), emotional well-being (consists of 6 items and ranging from 0 to 24, where higher scores indicating better quality of life). Each individual item was rated on a 5-point Likert scale, ranging from 0 (not at all good) to 4 (very well), where higher scores indicating better quality of life. FACT-G total score range was of 0 (not at all good) to 108 (very well), where higher scores indicating better quality of life.
Time Frame: as for outcome 37
Population: as for outcome 37
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 42
units on a scale
  Baseline | 80.22 [76.21 to 84.23]
  Change at Cycle 2: Day 1 | -1.15 [-4.10 to 1.80]
  Change at Cycle 3: Day 1: number analyzed (Participants) | 41
  Change at Cycle 3: Day 1 | -1.34 [-4.72 to 2.04]
  Change at Cycle 5: Day 1: number analyzed (Participants) | 38
  Change at Cycle 5: Day 1 | -0.36 [-3.21 to 2.48]
  Change at Cycle 7: Day 1: number analyzed (Participants) | 35
  Change at Cycle 7: Day 1 | -3.56 [-6.52 to -0.60]
  Change at Cycle 9: Day 1: number analyzed (Participants) | 35
  Change at Cycle 9: Day 1 | -2.39 [-4.94 to 0.16]
  Change at Cycle 11: Day 1: number analyzed (Participants) | 33
  Change at Cycle 11: Day 1 | -3.94 [-6.79 to -1.09]
  Change at Cycle 13: Day 1: number analyzed (Participants) | 29
  Change at Cycle 13: Day 1 | -4.74 [-8.11 to -1.37]
  Change at Cycle 15: Day 1: number analyzed (Participants) | 28
  Change at Cycle 15: Day 1 | -2.98 [-6.23 to 0.26]
  Change at Cycle 17: Day 1: number analyzed (Participants) | 28
  Change at Cycle 17: Day 1 | -4.64 [-7.37 to -1.91]
  Change at Cycle 19: Day 1: number analyzed (Participants) | 27
  Change at Cycle 19: Day 1 | -5.48 [-8.94 to -2.01]
  Change at Cycle 21: Day 1: number analyzed (Participants) | 27
  Change at Cycle 21: Day 1 | -4.34 [-7.94 to -0.74]
  Change at Cycle 23: Day 1: number analyzed (Participants) | 26
  Change at Cycle 23: Day 1 | -4.39 [-8.42 to -0.37]
  Change at Cycle 25: Day 1: number analyzed (Participants) | 24
  Change at Cycle 25: Day 1 | -3.22 [-6.94 to 0.50]
  Change at Cycle 27: Day 1: number analyzed (Participants) | 24
  Change at Cycle 27: Day 1 | -3.80 [-7.34 to -0.26]
  Change at Cycle 29: Day 1: number analyzed (Participants) | 23
  Change at Cycle 29: Day 1 | -4.52 [-8.58 to -0.45]
  Change at Cycle 31: Day 1: number analyzed (Participants) | 21
  Change at Cycle 31: Day 1 | -4.55 [-8.27 to -0.84]
  Change at Cycle 33: Day 1: number analyzed (Participants) | 20
  Change at Cycle 33: Day 1 | -6.67 [-10.26 to -3.08]
  Change at Cycle 35: Day 1: number analyzed (Participants) | 20
  Change at Cycle 35: Day 1 | -6.63 [-10.38 to -2.88]
  Change at Cycle 37: Day 1: number analyzed (Participants) | 19
  Change at Cycle 37: Day 1 | -6.49 [-10.52 to -2.46]
  Change at Cycle 39: Day 1: number analyzed (Participants) | 15
  Change at Cycle 39: Day 1 | -5.07 [-8.37 to -1.76]
  Change at Cycle 41: Day 1: number analyzed (Participants) | 11
  Change at Cycle 41: Day 1 | -5.06 [-9.92 to -0.20]
  Change at Cycle 43: Day 1: number analyzed (Participants) | 6
  Change at Cycle 43: Day 1 | -7.08 [-14.53 to 0.37]
  Change at Cycle 45: Day 1: number analyzed (Participants) | 3
  Change at Cycle 45: Day 1 | -5.94 [-27.36 to 15.47]
  Change at Cycle 47: Day 1: number analyzed (Participants) | 3
  Change at Cycle 47: Day 1 | -6.22 [-25.11 to 12.66]
  Change at Cycle 49: Day 1: number analyzed (Participants) | 2
  Change at Cycle 49: Day 1 | -8.58 [-90.11 to 72.95]
  End of Treatment: number analyzed (Participants) | 39
  End of Treatment | -7.09 [-10.98 to -3.20]

39. Secondary Outcome: Change From Baseline in Trial Outcome Index (TOI): Phase 2 at Day 1 of Cycle 2, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, 35, 37, 39, 41, 43, 45, 47, 49 and End of Treatment
Description: FACT is a modular approach to assess participant's health-related quality of life. TOI total score was derived from the sum of the 3 sub-scale scores: physical well-being, functional well-being (both sub-scales consisting of 7 items ranging from 0 to 28, where higher scores indicating better quality of life) and breast cancer subscale (consists of 9 items and ranging from 0 to 36, where higher scores indicating better quality of life). Each individual item was rated on a 5-point Likert scale, ranging from 0 (not at all good) to 4 (very well), where higher scores indicating better quality of life. TOI total score range was of 0 (not at all good) to 92 (very well), where higher scores indicating better quality of life.
Time Frame: as for outcome 37
Population: as for outcome 37
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 42
units on a scale
  Baseline | 71.52 [68.36 to 74.69]
  Change at Cycle 2: Day 1 | -1.17 [-3.24 to 0.89]
  Change at Cycle 3: Day 1: number analyzed (Participants) | 41
  Change at Cycle 3: Day 1 | -2.20 [-4.74 to 0.35]
  Change at Cycle 5: Day 1: number analyzed (Participants) | 38
  Change at Cycle 5: Day 1 | -2.54 [-5.25 to 0.16]
  Change at Cycle 7: Day 1: number analyzed (Participants) | 35
  Change at Cycle 7: Day 1 | -3.63 [-6.44 to -0.82]
  Change at Cycle 9: Day 1: number analyzed (Participants) | 35
  Change at Cycle 9: Day 1 | -3.31 [-6.03 to -0.60]
  Change at Cycle 11: Day 1: number analyzed (Participants) | 33
  Change at Cycle 11: Day 1 | -2.30 [-5.06 to 0.45]
  Change at Cycle 13: Day 1: number analyzed (Participants) | 29
  Change at Cycle 13: Day 1 | -3.93 [-7.31 to -0.56]
  Change at Cycle 15: Day 1: number analyzed (Participants) | 28
  Change at Cycle 15: Day 1 | -2.49 [-5.09 to 0.11]
  Change at Cycle 17: Day 1: number analyzed (Participants) | 28
  Change at Cycle 17: Day 1 | -3.18 [-6.02 to -0.34]
  Change at Cycle 19: Day 1: number analyzed (Participants) | 27
  Change at Cycle 19: Day 1 | -4.32 [-8.01 to -0.63]
  Change at Cycle 21: Day 1: number analyzed (Participants) | 27
  Change at Cycle 21: Day 1 | -3.56 [-6.83 to -0.28]
  Change at Cycle 23: Day 1: number analyzed (Participants) | 26
  Change at Cycle 23: Day 1 | -3.19 [-7.11 to 0.73]
  Change at Cycle 25: Day 1: number analyzed (Participants) | 24
  Change at Cycle 25: Day 1 | -2.13 [-5.51 to 1.26]
  Change at Cycle 27: Day 1: number analyzed (Participants) | 24
  Change at Cycle 27: Day 1 | -2.50 [-5.77 to 0.77]
  Change at Cycle 29: Day 1: number analyzed (Participants) | 23
  Change at Cycle 29: Day 1 | -3.70 [-7.36 to -0.03]
  Change at Cycle 31: Day 1: number analyzed (Participants) | 21
  Change at Cycle 31: Day 1 | -1.95 [-5.23 to 1.33]
  Change at Cycle 33: Day 1: number analyzed (Participants) | 20
  Change at Cycle 33: Day 1 | -4.30 [-7.65 to -0.95]
  Change at Cycle 35: Day 1: number analyzed (Participants) | 20
  Change at Cycle 35: Day 1 | -4.65 [-8.68 to -0.62]
  Change at Cycle 37: Day 1: number analyzed (Participants) | 19
  Change at Cycle 37: Day 1 | -4.84 [-8.77 to -0.92]
  Change at Cycle 39: Day 1: number analyzed (Participants) | 15
  Change at Cycle 39: Day 1 | -3.47 [-7.09 to 0.15]
  Change at Cycle 41: Day 1: number analyzed (Participants) | 11
  Change at Cycle 41: Day 1 | -2.27 [-7.62 to 3.08]
  Change at Cycle 43: Day 1: number analyzed (Participants) | 6
  Change at Cycle 43: Day 1 | -7.00 [-13.83 to -0.17]
  Change at Cycle 45: Day 1: number analyzed (Participants) | 3
  Change at Cycle 45: Day 1 | -3.00 [-22.40 to 16.40]
  Change at Cycle 47: Day 1: number analyzed (Participants) | 3
  Change at Cycle 47: Day 1 | -4.00 [-12.96 to 4.96]
  Change at Cycle 49: Day 1: number analyzed (Participants) | 2
  Change at Cycle 49: Day 1 | -2.00 [-14.71 to 10.71]
  End of Treatment: number analyzed (Participants) | 39
  End of Treatment | -6.03 [-9.61 to -2.45]

40. Secondary Outcome: Presence of Tumor Tissue Biomarker- Ki67: Phase 2
Description: Tumor tissue biomarker, Ki67 was analyzed to investigate possible associations with resistance or sensitivity to treatment with study drugs and was selected based on its known relevance to mechanisms involved in cell cycle regulation. Number of participants with less than or equal to and greater than 20 percent of Ki67 tumor tissue biomarker were reported.
Time Frame: Baseline (Day 1)
Population: Full analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991).
Measure: Number; unit: participants
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 42
participants
  <=20 percent | 19
  >20 percent | 23

41. Secondary Outcome: Presence of Tumor Tissue Biomarkers- Estrogen Receptor (ER) H-Score, Retinoblastoma (Rb) H-Score, B-cell Lymphoma-1 (BCL-1) H-Score, P16 H-Score: Phase 2
Description: Tumor tissue biomarkers ER, Rb, BCL-1 and P16 were analyzed to investigate possible associations with resistance or sensitivity to treatment with study drugs and were selected based on their known relevance to mechanisms involved in cell cycle regulation. Number of participants with positive ER (H-Score), Rb (H-Score), BCL-1 (H-Score) and P16 (H-Score) tumor tissue biomarkers were reported. The H-score is a method of assessing the extent of nuclear immunoreactivity, applicable to steroid receptors.
Time Frame: Baseline (Day 1)
Population: Full analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991).
Measure: Number; unit: participants
Arm/Group | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Number analyzed (Participants) | 42
participants
  ER (H-Score) | 41
  Rb (H-Score) | 41
  BCL-1 (H-Score) | 42
  P16 (H-Score) | 41

ADVERSE EVENTS:
Time Frame: Part 1 Phase 1: Lead-in period (Day -7) up to 28 days after last dose of study drug (up to 308 days), Part 2 Phase 1: Baseline (Day 1) up to 28 days after last dose of study drug (up to 1673 days), Phase 2: Baseline (Day 1) up to 28 days after last dose of study drug (up to 1526 days)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non serious in another participant, or 1 participant may have experienced both a serious and non serious event during the study. Safety analysis set included all enrolled participants who received at least 1 dose of study drug (PD-0332991).
Arm/Group | PD-0332991 100 mg: Dose Escalation Cohort | PD-0332991 125 mg: Dose Escalation Cohort | PD-0332991 125 mg+ Letrozole 2.5 mg: MTD Cohort | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 2/6 | 4/42
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PD-0332991 100 mg: Dose Escalation Cohort (N=6) | PD-0332991 125 mg: Dose Escalation Cohort (N=6) | PD-0332991 125 mg+ Letrozole 2.5 mg: MTD Cohort (N=6) | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort (N=42)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Malaise (General disorders) | 0 | 0 | 0 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PD-0332991 100 mg: Dose Escalation Cohort (N=6) | PD-0332991 125 mg: Dose Escalation Cohort (N=6) | PD-0332991 125 mg+ Letrozole 2.5 mg: MTD Cohort (N=6) | PD-0332991 125 mg+ Letrozole 2.5 mg: Expanded Cohort (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 10 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Constipation (Gastrointestinal disorders) | 1 | 2 | 2 | 12 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 9 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 1 | 32 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 5 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Malaise (General disorders) | 2 | 0 | 0 | 9 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2 | 19 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 6 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 9 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Alanine aminotransferase increased (Investigations) | 1 | 1 | 2 | 12 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 2 | 11 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Neutrophil count decreased (Investigations) | 5 | 4 | 6 | 34 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Platelet count decreased (Investigations) | 1 | 2 | 4 | 9 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Weight decreased (Investigations) | 1 | 1 | 1 | 5 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
White blood cell count decreased (Investigations) | 4 | 5 | 6 | 30 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 6 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 4 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Headache (Nervous system disorders) | 0 | 1 | 2 | 7 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 6 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 4 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 8 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 4 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 8 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Hypertension (Vascular disorders) | 0 | 0 | 1 | 5 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 5 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 9 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 5 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Influenza like illness (General disorders) | 0 | 0 | 0 | 5 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Angular cheilitis (Infections and infestations) | 0 | 0 | 0 | 4 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 4 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 4 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 3 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 8 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 3 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 4 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 4 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 4 | 5 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Pain (General disorders) | 0 | 0 | 0 | 3 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Pyrexia (General disorders) | 0 | 1 | 2 | 3 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 3 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 5 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 3 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 2 | 2 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Macular oedema (Eye disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 2 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Glossitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Fatigue (General disorders) | 0 | 2 | 2 | 2 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Mucosal inflammation (General disorders) | 0 | 0 | 2 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Influenza (Infections and infestations) | 0 | 0 | 1 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Blood creatinine increased (Investigations) | 2 | 0 | 1 | 2 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Parosmia (Nervous system disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 2 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Sensory disturbance (Nervous system disorders) | 0 | 0 | 1 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 3 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Cystitis (Infections and infestations) | 1 | 0 | 0 | 2 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Blood alkaline phosphatase increased (Investigations) | 2 | 2 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Lymphocyte count decreased (Investigations) | 1 | 3 | 0 | 2 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.
Genital haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 — MedDRA v17.1 was used for Dose Escalation Cohorts. MedDRA v20.1 was used for MTD Cohort. MedDRA v21.1 was used for Expanded Cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.